CLINICAL TRIAL: NCT00947869
Title: Glaucoma Including Pseudoexfoliation Syndrome (SFB 539)
Brief Title: Contrast Sensitivity in Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg (Other)
Responsible Party: University Eye Hospital Erlangen, University of Erlangen-Nürnberg
Organization: University of Erlangen-Nürnberg Medical School (Other)
Other Study IDs: DFG-SFB539-H
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Primary Open Angle Glaucoma; Secondary Open Angle Glaucoma Due to PEX
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The primary aim of the Erlangen´s Glaucoma Contrast Sensitivity-Study (EGCS-Study) is the evaluation of the diagnostic and prognostic validity of a diagnostic procedure, measuring contrast sensitivity. No therapeutic studies are performed.

ELIGIBILITY:
* Patients: Primary open angle glaucoma, secondary open angle glaucoma due to PEX
* Healthy volunteers (for reliability analysis)

Inclusion Criteria:

* Age > 18
* Best corrected visual acuity 0.8 or better
* European

Exclusion Criteria:

* eye diseases: Infantile glaucoma, angle glaucoma, secondary open angle glaucoma, wich are not due to PEX, diseases involving retina, condition after ophthalmological operations or trauma, cataract, diseases concerning the refractive system, age-related macular degeneration, diabetic retinopathy, optic neuropathy (MS, neuritis), amblyopia
* Any neurological diseases
* Systemic diseases with potentially ocular involvement (e.g., diabetes mellitus)
* Systemic drugs with potentially ocular involvement
* ocular drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-04

CONTACTS AND LOCATIONS:
Overall Officials: Anselm G Juenemann, Prof., Study Chair — University Erlangen-Nuremberg
Locations (1):
- University Eye Hospital, Erlangen, Bavaria, Germany